CLINICAL TRIAL: NCT05089344
Title: Growth Hormone Pretreatment in Poseidon Type IV Undergoing ICSI Using Minimal Induction Protocol: A Randomized Controlled Trial
Acronym: Growth hormone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed ElSaed Mostafa, principal investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH in poor responders
Record Dates: First submitted 2021-10-09; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Poor Response to Ovulation Induction Poseidon Type IV
MeSH Terms: interventions — Growth Hormone; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mild stimulation protocol + growth hormone adjuvant (Experimental): Controlled ovarian hyperstimulation protocol will be held according to a flexible GnRH antagonist protocol + Clomophine citrate.
  Ovarian stimulation will start with a fixed daily dose of 100 mg of Clomiphene citrate daily and recombinant FSH (Gonal-F®) will be started on day 2 of the menstrual cycle at a dose of 150 IU to be adjusted thereafter in a step up fashion every 2 to 4 days according to ovarian response .
  . For those in the GH group, 8 IU recombinant human GH will be administered starting from Day 14 of the previous cycle Till administration of HCG for ovulation triggering
  Interventions: Drug: Growth Hormone; Drug: Clomiphene citrate daily and recombinant FSH (Gonal-F®)
- Mild stimuation protocol (Active Comparator): Controlled ovarian hyperstimulation protocol will be held according to a flexible GnRH antagonist protocol + Clomophine citrate.
  Ovarian stimulation will start with a fixed daily dose of 100 mg of Clomiphene citrate daily and recombinant FSH (Gonal-F®) will be started on day 2 of the menstrual cycle at a dose of 150 IU to be adjusted thereafter in a step up fashion every 2 to 4 days according to ovarian response .
  .
  Interventions: Drug: Clomiphene citrate daily and recombinant FSH (Gonal-F®)

INTERVENTIONS:
Drug: Growth Hormone — growth hormone
  Arms: mild stimulation protocol + growth hormone adjuvant
Drug: Clomiphene citrate daily and recombinant FSH (Gonal-F®) — Clomiphene citrate daily and recombinant FSH (Gonal-F®)

SUMMARY:
This study is done aiming to Assess Efficiency of Growth hormone as an adjuvant in pretreatment of Poseidon type IV group " poor responders "undergoing ICSI using minimal induction protocol

DETAILED DESCRIPTION:
Patients are recruited from the attendee of the Infertility clinic and IVF unit in maternity hospital Ain shams university who are eligible for the trial.

Procedure will be done by Prof . Dr Mostafa Fouad . and Lecturer Dr Ebtihal ElTaieb

* Proper history taking, examination and investigations to:

* exclude other causes of infertility.
* Menstrual history: for assessment of oligo- or anovualtion.
* Medical history: .
* Past history: previous infertility treatment attempts or ovarian hyperstimulation syndrome.
* Obstetric history: for recurrent pregnancy loss.
* Clinical examination, including:
* Arterial blood pressure measurement
* Assessment of hirsutism via modified Ferriman-Gallwey score
* Assessment of alopecia and acne.
* Hormonal profile assessment: basal serum FSH, LH, E2, progesterone, AMH, total serum testosterone, SHBG (for calculation of FAI), DHEA, DHEAS, TSH, prolactin and 24-hour urinary free cortisol (to rule out Cushing's syndrome).
* Semen analysis: to rule out male cause of infertility as teratospermia or azospermia.
* Transvaginal ultrasonography: by the same experienced gynecological sonographer using a Voluson E6 Expert ultrasound machine (General Electric®, Fairfield, CT, USA) for U/S criteria of PCOS, AFC and exclusion any uterine or pelvic pathologies.
* Hysterosalpingography (HSG): to exclude any uterine, tubal or peritoneal abnormalities.

Patients fitting inclusion and exclusion criteria will be randomized to either study groups. A computer generated list via MedCalc ® Software, version 13.2.2 will be used, assigning each participant number to either study groups. Assignment will be done by sequentially numbered, otherwise identical, sealed envelopes (SNOSE), each containing a 2-inch by 2-inch paper with a written code designating the assigned group. These papers will be placed in a folded sheet of aluminum foil fitted inside the envelope. Effort will be taken to assure absence of any detectable differences in size or weight between intervention and control envelopes. Envelopes will be chosen to be opaque and lined inside with carbon paper. Envelopes will be opened sequentially only after writing the subject's tracking information on the envelope so that the carbon paper served as an audit trail.

After enrollment each patient randomly pick an envelope carrying a number, so that patients will not be aware of the assignment (single blind technique), then the controlled ovarian stimulation protocol will be applied according to letter enclosed (A or B) guided by the computer based randomization table.

The patients were randomly assigned to one of the two parallel groups:

* Group A: mild stimulation protocol + growth hormone adjuvant
* Group B: Mild stimulation protocol

Study Interventions: Patients in both groups received mild stimulation protocol:

Controlled ovarian hyperstimulation protocol will be held according to a flexible GnRH antagonist protocol + Clomophine citrate.

Ovarian stimulation will start with a fixed daily dose of 100 mg of Clomiphene citrate daily and recombinant FSH (Gonal-F®) will be started on day 2 of the menstrual cycle at a dose of 150 IU to be adjusted thereafter in a step up fashion every 2 to 4 days according to ovarian response (Kolibianakis et al., 2011).

. For those in the GH group, 8 IU recombinant human GH will be administered starting from Day 14 of the previous cycle Till administration of HCG for ovulation triggering, while those in the control group will receive the same stimulation protocol without the adjuvant GH treatment.

* Follow up TVU/S will be done every other day starting day 6 of stimulation.
* Cetrotide® 0.25 mg will be started when at least one of the following criteria is met: LH >10 IU/L, presence of a follicle with mean diameter >12 mm, and serum E2 level >150 pg/mL and continued until HCG administration.
* When the leading follicle reaches 16 mm, TV U/S will be performed daily till the largest follicle reach a diameter of >18mm. The maximum duration of rFSH stimulation will not be allowed to exceed day 16.
* OOCYTE RETRIEVAL, FERTILIZATION AND EMBRYO TRANSFER
* Ovarian pick up will be done 36 hours after HCG injection, the transducer will be connected to the ultrasound system. The direction of the guide beam will be checked. The puncturing needle will be connected to an aspiration apparatus attached by a fixation ring to the front and rear ends of the vaginal transducer, thereby defining the direction of puncture corresponding to the guide beam on the ultrasound image. Oocytes will be aspirated using the standard aspiration technique using Wallace® 101 catheter (Smiths medical®, Minnesota, USA) using aspiration pressure 90-100mmHg using flushing technique.

To maximize the number of oocytes recovered, follicular aspiration followed by a single 2-mL flush using embryo culture media. After initial aspiration, follicles were flushed and aspirated three times each with 2 mL flushing medium .

* Intracytoplasmic sperm injection will be performed on metaphase II oocytes using the direct penetration technique. Fertilization results will be assessed 16 to 19 hours after ICSI. Fertilization will be considered normal by the presence of two pronuclei. Oocyte degeneration was identified by collapse of cytoplamic contents and separation from the zona. Failed fertilization will be defined by the absence of the pronuclei.
* Embryo transfer will be performed on day 3 of ICSI, using ultrasound guidance in the midcorporeal part of the uterine cavity using soft Wallace® transfer catheter (Smiths medical®, Minnesota, USA).
* Luteal phase will be supported by natural progesterone in the form of vaginal suppositories 400 mg twice daily starting from the day of oocyte retrieval till pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* -Age group between 35 to 42 years old
* AFC <5
* AMH <1.2 ng/ml
* first IVF trial

Exclusion Criteria:

* - Serious and unstable disease, such as cerebrovascular, liver, and kidney disease "will be unfit for pregnancy".
* History of malignant or border line tumors "will be unfit for pregnancy".
* Endocrine or metabolic disorder "affecting quality of oocyte so affecting results".
* Either one of the couple with chromosomal abnormalities "affecting quality of oocyte so affecting results".
* Male partner with severe oligoasthenozoospermia or with teratozoospermia"affecting quality of embryo to be transfered so affecting results".
* Any contraindications to growth hormone, pregnancy (to be ruled out and documented before GH treatment).
* female patients with causes of infertility other than poor ovarian reserve
* females suffering from congenital or acquired uterine anomalies "will affect results of implantation and pregnancy rates "
* females with focal uterine lesions anomalies "will affect results of implantation and pregnancy rates "
* BMI >30 kg/m2 "affecting quality of oocyte so affecting results".

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 20 week of gestation
  pregnancy continuing after 20th week of gestation.

SECONDARY OUTCOMES:
- Biochemical pregnancy rate | 2 weeks after embryo transfer
  will be determined by positive pregnancy test performed 2 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Fouad, MD, Principal Investigator — Ainshams Maternity Hospital; Ebtihal ElTaieb, MD, Study Director — Ainshams Maternity Hospital
Locations (1):
- AinShams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No